CLINICAL TRIAL: NCT00309673
Title: Local Anesthesia Effect on Tuberculin Skin Test Results in Infants and Children
Brief Title: Local Anesthesia and Tuberculin Skin Test in Infants and Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CRC05001
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2006-04-03 (Estimated); Status verified 2006-03

CONDITIONS: Tuberculosis
Keywords: tuberculosis, tuberculin, childhood, pain
MeSH Terms: conditions — Tuberculosis; Pain | interventions — Lidocaine, Prilocaine Drug Combination

INTERVENTIONS:
Drug: lidocaine / Prilocaine

SUMMARY:
The use of local anaesthesia efficiently reduces pain due to needle puncture. However, when tuberculin skin test is performed it is the skin reaction to tuberculin injection that is studied. It is a quantitative skin reaction measured in millimiters. From the study of literature it is not known whether local anaesthetic modify skin reaction to tuberculin. Therefore, before recommending the use local anaesthesia for tuberculin intradermal injection we have to rule out a potential effect of local anaesthetic on the result of the test. This is particularly important in children, since there are more sensitive to pain than adults

ELIGIBILITY:
Inclusion Criteria:

hospitalized or non hospitalized infant or child (3 months-15 years)requiring a tuberculin skin test, in our hospital. hospitalized 1 to 3 months old infants requiring a tuberculin skin test, in our hospital.

-

Exclusion Criteria:

* child with contra indication to the use of Lidocaine / prilocaine
* child with evolutive dermatitis on forearms
* premature or newborn (less than 1 month of age)
* infants (1 - 24 months of age)who has yet received repeated local anaesthesia (at least 2)during the 24 previous hours
* infants (1 - 24 months of age)who is treated with a drug that could enhance the risk of methhaemoglobinemia
* child with previous evere local reaction to tuberculin injection (necrosis,ulceration)
* child with history of tuberculosis disease
* child with hepatic failure
* parents or the child himself if lod enough, have not given their agreement for the study

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60

PRIMARY OUTCOMES:
Measurement of tuberculin skin tests reaction performed with and without
local anaesthesia, in a child (intra subject reproducibility)

SECONDARY OUTCOMES:
influence of local anaesthesia use, on tuberculin skin test interpretation
between observer reproducibility
pain evaluation in child over 5 years of age between tuberculin skin tests performed with and without local anaesthesia
relationship between local anaesthesia use and failure to perform a correct intradermal injection
local tolerance to lidocaine / prilocaine

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Beydon, MD, Principal Investigator — APHP
Locations (1):
- Robert Debré Hospital, Paris, France